CLINICAL TRIAL: NCT03756350
Title: Clinical Evaluation of the Safety and Efficacy of a 1060nm Diode Laser for Non-invasive Fat Reduction of the Abdomen
Brief Title: Clinical Evaluation of the Safety and Efficacy of a 1060nm Diode Laser (Abdomen)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Venus Concept (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS1317
Record Dates: First submitted 2018-11-26; First posted 2018-11-28 (Actual); Results first posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-05

CONDITIONS: Fat Atrophy
Keywords: abdomen; adipose; fat
MeSH Terms: conditions — Platelet Glycoprotein IV Deficiency | interventions — Lasers, Semiconductor

STUDY DESIGN:
Masking Description: Blinded reviewer will evaluate the pre and post photos
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Treatment subjects (Experimental): Single group of subjects which will have the treatment of a 1060nm diode laser administered to them.
  Interventions: Device: 1060nm diode laser

INTERVENTIONS:
Device: 1060nm diode laser — Non-invasive medical aesthetic device designed for body contouring. The device is comprised of a console, four 1060nm diode laser applicators which are 60x60 mm in size. There is a belt included with the system to allow for the secure application of the applicators to the treatment area.

SUMMARY:
This study is evaluating a 1060nm diode laser for non-invasive fat reduction of the abdomen. The study will enrolled up to 50 subjects requesting non-invasive lipolysis of the abdomen. Each subject will receive a single study treatment. Subjects will be followed at six and twelve weeks post treatment. Twelve week outcomes will be compared to baseline.

DETAILED DESCRIPTION:
Open-label baseline controlled evaluator-blind multi-centre study evaluating a 1060nm diode laser for non-invasive fat reduction of the abdomen. The study will enrolled up to 50 subjects requesting non-invasive lipolysis of the abdomen. Each subject will receive a single study treatment which takes approximately 25 minutes. Subjects will be followed at six and twelve weeks post treatment. Twelve week outcomes will be compared to baseline.

ELIGIBILITY:
Inclusion Criteria:

* able to read, understand and voluntarily provide written informed consent
* healthy male or female > 18 years of age seeking treatment for unwanted fat in the abdomen
* BMI score is less then 30
* agree to not making any major changes in their diet or lifestyle during the course of the study
* able and willing to comply with the treatment / follow up schedule and requirements
* women of child-bearing age are required to be using a reliable method of birth control at least 3 months prior to study enrolment and for the duration of the study, have a negative urine pregnancy test baseline

Exclusion Criteria:

* pregnant in the last 3 months intending to become pregnant, postpartum or nursing in the last 6 months
* any previous liposuction / lipo-sculpture or any type of surgical procedure in the treatment area in the past 12 months
* history of immunosuppression / immune deficiency disorders including AIDS and HIV infection, or use of immunosuppressive medications, 6 month prior to and during the course of the study
* History of hyperlipidemia, diabetes, hepatitis, blood coagulopathy or excessive bleeding
* Use of antiplatelet medications (81 mg of acetylsalicylic acid daily is permitted), anticoagulants, thrombocytes or any-inflammatory medications within 2 weeks of treatment
* Having a history of skin cancer or any other cancer in the area to be treated, including presence of malignant or pre-malignant pigmented lesions
* Having a permanent implant in the treatment area such as a metal plate or injected chemical substance such as silicone pr parenteral gold therapy (gold sodium thiomalate)
* Use of medications, herbs or food supplements and vitamins known to induce photosensitivity to light exposure at the wavelength used history of photosensitivity disorder
* Suffering from significant skin conditions in the treatment area or inflammatory skin conditions including but not limited to open lacerations, abrasions, herpes sores, cold sores, active infections
* Tattoos in the treatment area
* Poor quality skin (laxity)
* Abdominal wall, muscular abnormality or hernia on physical examination
* Unstable weight within the last 6 months (+ or - 3% weight change in the prior six months)
* Participation in another clinical study involving the same anatomical areas within the last 6 months
* History of keloid and hypertrophic scar formation or poor wound healing in the treatment area
* As per the investigators discretion any physician or mental condition which may make it unsafe for the subject to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-11-14 (Actual); Primary Completion 2019-07-02 (Actual); Study Completion 2019-07-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Kilmer, MD, Principal Investigator — Skin and Laser Surgery Center of Northern California; Jeffery Kenkel, MD, Principal Investigator — UT Southwestern
Locations (2):
- United States (2):
  - Laser and Skin Surgery Center of Northern California, Sacramento, California
  - Southwestern Medical Center Department of Plastic Surgery, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Decorato JW, Chen B, Sierra R. Subcutaneous adipose tissue response to a non-invasive hyperthermic treatment using a 1,060 nm laser. Lasers Surg Med. 2017 Jul;49(5):480-489. doi: 10.1002/lsm.22625. Epub 2017 Jan 19. PMID 28103642
- [Result] Katz B, Doherty S. Safety and Efficacy of a Noninvasive 1,060-nm Diode Laser for Fat Reduction of the Flanks. Dermatol Surg. 2018 Mar;44(3):388-396. doi: 10.1097/DSS.0000000000001298. PMID 28902034
- [Result] McBean JC, Katz BE. Laser lipolysis: an update. J Clin Aesthet Dermatol. 2011 Jul;4(7):25-34. No abstract available. PMID 21779417
- [Result] Schilling L, Saedi N, Weiss R. 1060 nm Diode Hyperthermic Laser Lipolysis:The Latest in Non-Invasive Body Contouring. J Drugs Dermatol. 2017 Jan 1;16(1):48-52. PMID 28095532

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment Subjects
Started | 30
Completed | 29
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment Subjects
Number analyzed (Participants) | 29
Age, Continuous [Mean (Full Range); unit: years] | 45 [26 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 2
  White | 22
  More than one race | 2
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Before and After Photograph Sets Correctly Identified by Independent, Blinded Evaluators
Description: Photographic evaluation by independent blinded evaluators with correct identification of pre-treatment baseline images when compared to post-treatment images taken at 12 weeks
Time Frame: Week 12 vs baseline
Population: All subjects who had baseline and Week 12 follow up photos.
Measure: Number; unit: Photo sets
Units Other Than Participants: Photo sets
Arm/Group | Treatment Subjects
Number analyzed (Participants) | 27
Number analyzed (Photo sets) | 81
Photo sets | 54

2. Secondary Outcome: Change in Fat Thickness
Description: Change in thickness of the adipose layer as measured by ultrasound at 12 weeks post-treatment as compared to baseline
Time Frame: week 12
Measure: Median (Standard Error); unit: Percent change in abdominal fat
Arm/Group | Treatment Subjects
Number analyzed (Participants) | 29
Percent change in abdominal fat | -9.8 (1.56)

3. Secondary Outcome: Subject Satisfaction
Description: Subject satisfaction with treatment at 12 weeks after treatment using the 5-point Likert Subject Satisfaction Scale. A score of 4 is very satisfied and 0 is very unsatisfied.
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Subjects
Number analyzed (Participants) | 29
score on a scale | 2.9 (0.85)

4. Secondary Outcome: Treatment Pain
Description: Subject assessment of discomfort and pain post treatment as measured using the Wong Baker Faces Scale, which is a 10 point scale with 10 being the worst pain ever and 0 being no pain.
Time Frame: Week 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Subjects
Number analyzed (Participants) | 29
score on a scale | 2.6 (1.6)

ADVERSE EVENTS:
Time Frame: 12 weeks following treatment
Arm/Group | Treatment Subjects
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 2/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Subjects (N=30)
Not visible, but palpable nodules (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-19): https://cdn.clinicaltrials.gov/large-docs/50/NCT03756350/Prot_SAP_000.pdf